CLINICAL TRIAL: NCT02953353
Title: Noninvasive Neuromodulation of the Prefrontal Cortex in Subjects With Obesity: a Proof-of-concept Study
Brief Title: Noninvasive Neuromodulation of the Prefrontal Cortex in Subjects With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Beth Israel Deaconess Medical Center (Other); USDA Human Nutrition Research Center on Aging (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vivian Marques Miguel Suen, Professor of Internal Medicine Department at Ribeirão Preto, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Process HCRP: 8463/2016
Record Dates: First submitted 2016-10-17; First posted 2016-11-02 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Obesity; Feeding behavior; Transcranial direct current stimulation; Weight loss
MeSH Terms: conditions — Obesity; Feeding Behavior; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active group (Active Comparator): Active transcranial direct current stimulation (tDCS) and hypocaloric diet.
  Interventions: Device: Active transcranial direct current stimulation (tDCS); Other: Hypocaloric diet
- Control group (Sham Comparator): Sham transcranial direct current stimulation (tDCS) and hypocaloric diet.
  Interventions: Other: Hypocaloric diet; Other: Sham transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Active transcranial direct current stimulation (tDCS) — Participants will receive 10 daily sessions (phase 2) and 3 times a week (phase 3) of tDCS (2mA, 30 min per session). The tDCS montage will target the left dorsolateral prefrontal cortex (DLPFC) (anode: F3 based on the 10:20 system; cathode over the right supraorbital area). For stimulation the investigators will use 5x5cm sponge pads that will be soaked in 0.9% saline during the sessions.
  Arms: Active group
Other: Hypocaloric diet — During phase 3, participants will undergo a supervised hypocaloric diet intervention for 2 weeks based on a low-calorie diet (LCD) providing a hypocaloric diet based in 20% reduction from total energy expenditure (TEE). The diet will be individualized on the basis of physical activity levels, age for each participant. This intervention will be be conducted at an inpatient, well-controlled setting to guarantee adherence to the diet. Here the diet intervention will be administered in combination with tDCS. tDCS will be applied every other day (Monday, Wednesday, Friday) over the course of these two weeks.
Other: Sham transcranial direct current stimulation (tDCS) — Subjects in the control group will receive sham stimulation (placebo) (similar procedure and duration as real tDCS, but here electric current flows for 30 s only, to mimic the subjective sensations that occur with active tDCS).
  Arms: Control group

SUMMARY:
The overall goal of this proposal is to evaluate the efficacy of transcranial direct current stimulation (tDCS), a noninvasive neuromodulation technique, to facilitate weight loss and weight loss maintenance in obesity. This is a novel clinical research study that examines the therapeutic potential of an innovative biomedical treatment for weight loss.

DETAILED DESCRIPTION:
The hypothesis is that tDCS will successfully engage prefrontal-related neurobehavioral cognitive control systems, resulting in decreased eating disinhibition and therefore facilitation of weight loss and weight loss maintenance. To test this hypothesis, a 6-month randomized, sham-controlled, double-blind, intervention study was designed. Subjects will undergo an intervention with the following components/phases:

1. Phase 1 - Target engagement (one session) The purpose of this phase is to examine whether tDCS can reach the brain target, the dorsolateral prefrontal cortex, and influence performance in a neuropsychology tests that depends on the activity of this region. Results from this component of the study will provide evidence for target engagement. Genomic DNA will be extracted from whole blood for sequencing of Catechol-O-methyltransferase (COMT) and brain-derived neurotrophic factor (BDNF) polymorphism genotypes.
2. Phase 2 - tDCS alone (two weeks) During this phase participants will receive daily tDCS sessions over the course of two weeks (Monday to Friday; total=10 sessions). The purpose of this phase is to examine the effect of modulating the activity of the prefrontal cortex with tDCS on body weight under baseline/weight stable conditions. Also analyse changes in appetite and eating behavior.
3. Phase 3 - tDCS plus hypocaloric diet (two weeks). During this phase participants will undergo a hypocaloric diet intervention aimed at achieving a 5% body weight reduction at 3 months. The diet will be individualized on the basis of physical activity levels, age for each participant. This intervention will be be conducted at an inpatient, well-controlled setting to guarantee adherence to the diet. Here the diet intervention will be administered in combination with tDCS. tDCS will be applied every other day (Monday, Wednesday, Friday) over the course of these two weeks. The purpose of this component is to examine acute changes in weight associated with tDCS in combination with the diet. Also analyse changes in appetite and eating behavior.
4. Phase 4 - Follow up (6 months). During this phase (outpatient) changes in body weight over time will be assessed to evaluate weight maintenance. Subjects will be asked to come back to the laboratory at 1, 3 and 6 months. Also analyse changes in appetite and eating behavior.

ELIGIBILITY:
Inclusion Criteria:

* Women with obesity (BMI 30-35 kg/m2), with stable weight over the previous 3 months.

Exclusion Criteria:

* pregnancy
* diabetes
* acute and chronic kidney disease
* pancreatitis
* any active psychiatric or neurological condition at the time of joining the study
* intake of centrally-acting medications that could interfere with tDCS effects
* anemia (Hgb <12 g/dl)
* any other significant medical condition
* contraindications for tDCS, which includes damaged skin at the site of stimulation, any electrically sensitive or metallic device and history of epilepsy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 months
  The primary outcome will be change in body weight after two weeks intervention (tDCS alone) versus baseline (day 1), the change in body weight between the beginning and the end of the inpatient period (tDCS plus hypocaloric diet), and the change in body weight throughout follow-up (6 months), i.e. between the end of the tDCS intervention (end of the inpatient phase) and the end of the study.

SECONDARY OUTCOMES:
Appetite visual analogue scale | 6 months
  The investigators will analyse changes in appetite during the different phases of the study: phase 1 (target engagement), phase 2 (tDCS-only effect), phase 3 (tDCS plus diet effect), phase 4 (follow-up) using the visual analogue scale.
Eating behavior questionnaire | 6 months
  The investigators will analyse changes in eating behavior during the different phases of the study: phase 1 (target engagement), phase 2 (tDCS-only effect), phase 3 (tDCS plus diet effect), phase 4 (follow-up) using the three-factor eating and food craving questionnaires.
Cognitive performance in a food modified working memory test | 2 weeks
  The investigators will compare accuracy and reaction times before and after the 2 weeks with tDCS only. To evaluate working memory performance an N-back task will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian MM Suen, MD PhD, Principal Investigator — University of Sao Paulo; Sai K Das, PhD, Principal Investigator — Human Nutrition Research Center on Aging, Tufts University; Miguel Alonso-Alonso, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (3):
- United States (2):
  - Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
- Clinical Hospital of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] CREUTZFELDT OD, FROMM GH, KAPP H. Influence of transcortical d-c currents on cortical neuronal activity. Exp Neurol. 1962 Jun;5:436-52. doi: 10.1016/0014-4886(62)90056-0. No abstract available. PMID 13882165
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Okamoto M, Dan H, Sakamoto K, Takeo K, Shimizu K, Kohno S, Oda I, Isobe S, Suzuki T, Kohyama K, Dan I. Three-dimensional probabilistic anatomical cranio-cerebral correlation via the international 10-20 system oriented for transcranial functional brain mapping. Neuroimage. 2004 Jan;21(1):99-111. doi: 10.1016/j.neuroimage.2003.08.026. PMID 14741647
- [Background] Truong DQ, Magerowski G, Blackburn GL, Bikson M, Alonso-Alonso M. Computational modeling of transcranial direct current stimulation (tDCS) in obesity: Impact of head fat and dose guidelines. Neuroimage Clin. 2013 May 31;2:759-66. doi: 10.1016/j.nicl.2013.05.011. eCollection 2013. PMID 24159560
- [Background] Truong DQ, Magerowski G, Pascual-Leone A, Alonso-Alonso M, Bikson M. Finite Element study of skin and fat delineation in an obese subject for transcranial Direct Current Stimulation. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:6587-90. doi: 10.1109/EMBC.2012.6347504. PMID 23367439
- [Background] Alonso-Alonso M. Translating tDCS into the field of obesity: mechanism-driven approaches. Front Hum Neurosci. 2013 Aug 27;7:512. doi: 10.3389/fnhum.2013.00512. eCollection 2013. PMID 23986687
- [Background] Gluck ME, Alonso-Alonso M, Piaggi P, Weise CM, Jumpertz-von Schwartzenberg R, Reinhardt M, Wassermann EM, Venti CA, Votruba SB, Krakoff J. Neuromodulation targeted to the prefrontal cortex induces changes in energy intake and weight loss in obesity. Obesity (Silver Spring). 2015 Nov;23(11):2149-56. doi: 10.1002/oby.21313. PMID 26530931
- [Background] Val-Laillet D, Aarts E, Weber B, Ferrari M, Quaresima V, Stoeckel LE, Alonso-Alonso M, Audette M, Malbert CH, Stice E. Neuroimaging and neuromodulation approaches to study eating behavior and prevent and treat eating disorders and obesity. Neuroimage Clin. 2015 Mar 24;8:1-31. doi: 10.1016/j.nicl.2015.03.016. eCollection 2015. PMID 26110109